CLINICAL TRIAL: NCT06869551
Title: A Phase 3, Multicenter, Double-blind, Placebo-controlled, Randomized Withdrawal Trial to Evaluate the Efficacy, Safety, and Pharmacokinetics of Deucravacitinib in Children and Adolescents From 5 to Less Than 18 Years of Age With Active Juvenile Psoriatic Arthritis
Brief Title: A Study to Evaluate the Drug Levels, Efficacy, and Safety of Deucravacitinib (BMS-986165) in Pediatric Participants With Juvenile Psoriatic Arthritis
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IM011-1071
Record Dates: First submitted 2025-03-06; First posted 2025-03-11 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Juvenile Psoriatic Arthritis
Keywords: Juvenile Psoriatic Arthritis (JPsA); Juvenile Idiopathic Arthritis (JIA); Pediatric PsA; Deucravacitinib; BMS-986165
MeSH Terms: conditions — Arthritis, Juvenile | interventions — deucravacitinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental)
  Interventions: Drug: Deucravacitinib
- Arm B (Placebo Comparator)
  Interventions: Drug: Deucravacitinib; Other: Placebo

INTERVENTIONS:
Drug: Deucravacitinib — Specified dose on specified days
Other: Placebo — Specified dose on specified days
  Arms: Arm B

SUMMARY:
The purpose of this study is to evaluate the drug levels, efficacy, and safety of Deucravacitinib (BMS-986165) in pediatric participants with juvenile psoriatic arthritis.

ELIGIBILITY:
Inclusion Criteria

* Participants must have been diagnosed with Juvenile Psoriatic Arthritis (JPsA).
* Participants must have at least three joints that are affected by arthritis.
* Participants must have tried at least one type of medicine for JPsA for at least three months, but it didn't work well or caused problems.

Exclusion Criteria

* Participants must not have been diagnosed with JPsA before 5 years of age.
* Participants must not have other types of Juvenile Idiopathic Arthritis (JIA) that aren't JPsA,
* Participants must not have a history of chronic eye inflammation (uveitis), or were diagnosed with uveitis within the last three months.
* Other protocol-defined Inclusion/Exclusion criteria apply.

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2025-03-13 (Actual); Primary Completion 2030-03-06 (Estimated); Study Completion 2031-03-04 (Estimated)

PRIMARY OUTCOMES:
Time to first flare during the withdrawal period | From week 16 up to week 42

SECONDARY OUTCOMES:
Trough concentration at steady state (Cminss) | At week 16
Time-averaged steady-state concentration (Cavgss) | At week 16
Steady-state maximum observed concentration (Cmaxss) | At week 16
Number of participants with flare during the withdrawal period | From week 16 up to week 42
Number of participants achieving each of American College of Rheumatology (ACR) Pedi (30/50/70/90) | At week 16 and week 42
Change from baseline in juvenile idiopathic arthritis-American College of Rheumatology (JIA-ACR) Pedi Core Criteria | At week 16 and week 42
Number of participants achieving low disease activity (Juvenile arthritis disease activity 71-joint score based on C-reactive protein (JADAS71-CRP) score: for oligoarthritis 1.1 to 2; for polyarthritis 1.1 to 3.8) | At week 16 and week 42
Number of participants achieving inactive disease (JADAS71-CRP score ≤ 1) | At week 16 and week 42
Number of participants attaining clinical remission for at least 6 consecutive months | At week 42
Number of participants achieving psoriasis area and severity index (PASI) 75 | At week 42
Number of participants for each assessment who evaluate palatability scale as ≥ 3 (good or better), swallowability scale as ≤ 4 (neutral or easier), and taste scales (Sweetness, Bitterness, Flavor, and Overall Taste) as "None" or "Weak" | At week 16
Assessment of exposure-response (E-R) utilizing steady-state exposure of deucravacitinib from the pharmacokinetic (PK) analysis and efficacy results using ACR Pedi 30 | At week 16
Number of participants with adverse events (AEs) | Up to week 42
Number of participants with adverse event of special interest (AESIs) | Up to week 42
Number of participants with AEs leading to discontinuation | Up to week 42
Number of participants with serious adverse events (SAEs) | Up to week 42
Number of participants with Uveitis | Up to week 42

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (46):
- United States (7):
  - Local Institution - 0038, Lancaster, California
  - Local Institution - 0020, Chicago, Illinois
  - Local Institution - 0023, Indianapolis, Indiana
  - Local Institution - 0059, North New Hyde Park, New York
  - Local Institution - 0065, Cincinnati, Ohio
  - Local Institution - 0066, Cleveland, Ohio
  - Local Institution - 0036, Austin, Texas
- Brazil (13):
  - Local Institution - 0068, Fortaleza, Ceará
  - Local Institution - 0032, Cuiabá, Mato Grosso
  - Local Institution - 0030, Belo Horizonte, Minas Gerais
  - Local Institution - 0013, Curitiba, Paraná
  - Local Institution - 0072, Curitiba, Paraná
  - Local Institution - 0007, Recife, Pernambuco
  - Local Institution - 0033, Porto Alegre, Rio Grande do Sul
  - Local Institution - 0008, Porto Alegre, Rio Grande do Sul
  - Local Institution - 0069, Xangri-lá, Rio Grande do Sul
  - Local Institution - 0073, Vila Clementino, São Paulo-SP
  - Local Institution - 0027, Rio de Janeiro
  - Local Institution - 0047, São Paulo
  - Local Institution - 0010, São Paulo
- Bulgaria (2):
  - University Multiprofile Hospital for Active Treatment "Sveti Georgi" EAD, Plovdiv
  - Local Institution - 0062, Sofia
- China (7):
  - Local Institution - 0049, Beijing, Beijing Municipality
  - The Children's Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Local Institution - 0060, Guangzhou, Guangdong
  - Childrens Hospital of Nanjing Medical University, Nanjing, Jiangsu
  - The First Hospital of Jilin University, Changchun, Jilin
  - The Children's Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Children's Hospital of Fudan University, Shanghai
- Czechia (2):
  - Fakultni nemocnice Olomouc, Olomouc, Olomoucký kraj
  - Fakultni nemocnice v Motole, Prague, Praha 5
- Germany (2):
  - Kinderklinik des Uni-Klinikums Erlangen, Erlangen
  - Praxis Kinder- und Jugendrheumatologie Dr. Ivan Foeldvari, Hamburg
- Italy (2):
  - University of Naples Federico II, Napoli, Campania
  - Azienda Ospedaliera Universitaria Meyer IRCCS, Florence, Tuscany
- Local Institution - 0017, San Juan, Puerto Rico
- Romania (3):
  - Spitalul Clinic de Urgenta pentru Copii Cluj-Napoca, Cluj-Napoca, Cluj
  - Local Institution - 0048, Iași, Iaşi
  - Sc Medaudio-Optica Srl, Râmnicu Vâlcea, Vâlcea County
- Spain (3):
  - Hospital Universitari Vall d'Hebron, Barcelona, Barcelona [Barcelona]
  - Hospital Universitario Ramón y Cajal, Madrid, Madrid, Comunidad de
  - Hospital Universitari i Politecnic La Fe, Valencia
- Turkey (Türkiye) (4):
  - Istanbul Universitesi Cerrahpasa, Istanbul- Fatih, Istanbul
  - Local Institution - 0061, Ankara
  - Local Institution - 0044, Ankara
  - Umraniye Training and Research Hospital, Istanbul

IPD SHARING:
Plan to Share IPD: Yes
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria. Additional information regarding Bristol Myer Squibb's data sharing policy and process can be found at: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosure-commitment.html
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See plan description
Access Criteria: See plan description
URL: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosure-commitment.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsclinicaltrials.com/us/en/clinical-trials/NCT06869551.html